CLINICAL TRIAL: NCT05743101
Title: Safety and Efficacy Study of Levofloxacin Combined With Endovascular Thrombectomy for Acute Ischemic Stroke Due to Large Vessel Occlusion of Anterior Circulation
Brief Title: Safety and Efficacy Study of Levofloxacin Combined With Endovascular Thrombectomy for Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVX-EVT
Record Dates: First submitted 2023-02-06; First posted 2023-02-24 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Endovascular thrombectomy, Levofloxacin
MeSH Terms: conditions — Ischemic Stroke | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levofloxacin group (Experimental): Levofloxacin 200mg twice per day is administrated.
  Interventions: Drug: Levofloxacin
- Levofloxacin simulant group (Placebo Comparator): Levofloxacin simulant 200mg twice per day is administrated.
  Interventions: Drug: Levofloxacin simulant

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin is a quinolone antibiotics and newly identified neuro-protective agent.Endovascular thrombectomy is one of the treatments for acute ischemic stroke.
  Other Names: Endovascular thrombectomy
  Arms: Levofloxacin group
Drug: Levofloxacin simulant — Levofloxacin simulant is placebo.Endovascular thrombectomy is one of the treatments for acute ischemic stroke.
  Other Names: Endovascular thrombectomy
  Arms: Levofloxacin simulant group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of levofloxacin combined with endovascular thrombectomy in treating acute ischemic stroke due to large vessel occlusion of anterior circulation.

DETAILED DESCRIPTION:
Acute ischemic stroke is a leading cause of disability and mortality. Emergency thrombectomy is the highest recommended treatment for patients with large vessel occlusion. However, there are still some patients with severe disability or mortality within 90 days after surgery. It is necessary to find new interventions combined to endovascular thrombectomy, which promote the efficacy of endovascular thrombectomy. The investigators' previous studies suggested levofloxacin to be a newly identified neuro-protective agent, which could reduce infarct volume and improve neurologic function in animal models.To evaluate the efficacy and safety of levofloxacin combined with endovascular thrombectomy in treating acute ischemic stroke patients due to large vessel occlusion of anterior circulation, the prospective, multicenter and randomized controlled trial was designed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Patients with clinically confirmed acute ischemic stroke within 24 hours after onset, CTA or DSA confirmed anterior circulation large vessel occlusion (ICA, M1/proximal M2 segment of MCA, tandem lesions), met the current guidelines for emergency endovascular interventional therapy, and underwent emergency thrombectomy.
3. mRS≤1 before stroke onset.
4. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Patients with contraindications to emergency thrombectomy;
2. The head CT showed large facial cerebral infarction;
3. Patients using glucocorticoids, antiarrhythmic drugs (class I and class III antiarrhythmic drugs: quinidine, procaine amine, lidocaine, phenytoin sodium, verapamil, etc.), and quinolones within 14 days;
4. Patients with other diseases that may aggravate adverse drug reactions, such as ventricular arrhythmias, prolonged QT interval (male: QTc>430ms, female: QTc>450ms), severe cardiac insufficiency (NYHA functional grade ≥ III), myasthenia gravis, peripheral neuropathy, seizures, tendon-related diseases, severe immune system-related diseases, hematological diseases, active hepatitis or cirrhosis, serious respiratory diseases;
5. Abnormal liver and kidney function: glutamic oxaloacetic transaminase or glutamic pyruvic transaminase exceeds 3 times the upper limit of normal; Direct bilirubin or indirect bilirubin more than 3 times the normal upper limit; Blood creatinine exceeds 1.1 times the upper limit of normal; Creatinine clearance rate≤50ml/min; Urea nitrogen≥ 20mg/dL;
6. Fasting blood glucose lower than 3.9 mmol/L;
7. Patients allergy to fluoroquinolones or other antibiotics;
8. Patients with a life expectancy less than 3 months or patients unable to complete the study for other reasons;
9. Not willing to be followed up or poor treatment compliance;
10. Patients who are participating in other clinical studies, or have participated in other clinical studies within 3 months before enrollment, or have participated in this study;
11. Other conditions not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) after 3 days of Levofloxacin/simulant treatment | immediately after 3 days of Levofloxacin/simulant treatment
  National Institute of Health stroke scale (NIHSS) ranged from 0 to 42, a low value represents a better outcome.
NIHSS at discharge/7 days | discharge/7 days
  National Institute of Health stroke scale (NIHSS) ranged from 0 to 42, a low value represents a better outcome.

SECONDARY OUTCOMES:
Hemorrhagic transformation and symptomatic intracranial hemorrhage | 24h,3days and discharge/7 days
  defined by computed Tomography (CT) brain scan suggested bleeding, accompanied by an increase in National Institute of Health stroke scale (NIHSS) score of ≥4 points.
Infarct volume after 3 days of Levofloxacin/simulant treatment | immediately after 3 days of Levofloxacin/simulant treatment
  assessed by magnetic resonance imaging brain scan
Modified rankin scale (mRS) score at 30 days | 30 days
  Modified Rankin Scale (mRS), ranged from 0 to 6, a low value represents a better outcome.
mRS score at 90 days | 90 days
  Modified Rankin Scale (mRS), ranged from 0 to 6, a low value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD,PhD, Principal Investigator — The First Hospital of Jilin University